CLINICAL TRIAL: NCT01920594
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind (Sponsor Open) Study of GSK1278863, a HIF-Prolyl Hydroxylase Inhibitor, to Reduce Ischemic Events in Patients Undergoing Thoracic Aortic Aneurysm Repair
Brief Title: Study of GSK1278863 to Reduce Ischemic Events in Patients Undergoing Thoracic Aortic Aneurysm Repair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116097
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Surgical Procedures
Keywords: GSK1278863; Thoracic Aortic Aneurysm Repair
MeSH Terms: interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GSK1278863 (Experimental): Subject will receive GSK1278863 300mg on Day-1 (12 +/- 4 hours prior to planned surgery) as a loading dose followed by GSK1278863 100mg once daily for 4 days starting from Day 0.
  Interventions: Drug: GSK1278863
- Placebo (Placebo Comparator): Subject will receive GSK1278863 matching placebo on Day-1 (12 +/- 4 hours prior to planned surgery) as a loading dose followed by GSK1278863 matching placebo once daily for 4 days starting from Day 0.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1278863 — White, round biconvex, film coated tablet with unit dose strength of 100 mg for oral administration
  Arms: GSK1278863
Drug: Placebo — White, round biconvex, film coated GSK1278863 matching placebo tablet for oral administration
  Arms: Placebo

SUMMARY:
This study will test the hypothesis that GSK1278863 will reduce neurologic, renal, and/or cardiac ischemia in patients undergoing elective descending thoracic aorta/thoracoabdominal aortic aneurysm (DTA/TAAA) repair, a population known to be at high risk for ischemic events from their underlying pathology and the surgical complexity required to address their disease. Approximately 160 subjects will be stratified according to intervention type (surgical or endovascular repair, with the latter limited to 50% of the total study population) and randomized in a 1:1 fashion to treatment with GSK1278863 (300 milligrams [loading dose] followed by 100 milligrams [mg]/day x 4 days) or placebo starting prior to planned repair, through postoperative day 3. The duration of participation in this study is expected to be approximately 4 to 8 weeks from screening to follow-up.

ELIGIBILITY:
Inclusion Criteria

* Adults >= 18 years of age who require the following types of descending thoracic aorta or thoracoabdominal aorta repair for atherosclerotic aneurysm or chronic dissection (de novo Type B or residual Type B [following Type A repair]) via open surgery or endovascular stenting (TEVAR) as per their treating surgeon
* Open surgery:

Extent I TAAA (+/-distal arch) if it extends to or beyond renal ostia. Extent II TAAA (+/-distal arch). Extent III TAAA (defined as proximal extent or anastamosis superior to inferior pulmonary vein).

Extent IV TAAA only with a prior TEVAR or if it is a redo procedure (in this setting a "redo" is a prior abdominal aortic aneurysm (AAA) open or endovascular aortic repair (EVAR), with either proximal suture line disruption or mesenteric segment aneurysm recurrence requiring redo Extent IV reconstruction).

DTA repair with one of the following: Safi extent C coverage. Subclavian to diaphragm disease extent. >75% of total DTA length.

-TEVAR with one of the following: Full DTA coverage with previous abdominal EVAR or open AAA. Full DTA coverage including Zone 2 to celiac (i.e., distal arch plus full coverage DTA).

Full DTA coverage with celiac artery coverage with or without left subclavian artery coverage (Zone 2 or Zone 3 proximal landing), or full DTA (either Zone 2 or Zone 3) with extension distal to celiac with visceral debranching (e.g., the abdominal hybrid Extent 2 TAAA).

Note: Zone 2 is defined as between the left carotid through coverage of the left subclavian artery and Zone 3 is defined as the first 3cm distal to the left subclavian (e.g., between left subclavian and ligamentum [isthmus]).

* Completed any staging or bypass procedure that precedes the aortic repair at least 48 hours prior to the repair.
* Expect placement of a lumbar CSF catheter during the procedure with plans to maintain it for at least 48 hours per the treating physician.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli international unit /mililiter (mL) and estradiol < 40 picogram/mL (<147 picomoles/Liter) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Child-bearing potential and agrees to use one of the contraception methods from screening until completion of the Follow-up Visit.

* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of Screening until the completion of the Follow-up Visit.

Exclusion Criteria

* The subject has a traumatic aortic dissection.
* The subject has a baseline NIHSS > 1 or modified Rankin Scale > 1.
* The subject has a history of myocardial infarction, stroke, or spinal infarct within the past 3 months.
* The subject has active ulcer disease or recent gastrointestinal bleeding within the past 6 months.
* The subject has a history of deep venous thrombosis or pulmonary embolism in the past 12 months.
* The subject has been treated for a malignancy (excluding non-melanomatous skin cancers) within the past 12 months and is not confirmed to be disease free.
* The subject has had treatment for retinal neovascularization (e.g., diabetic proliferative retinopathy or age related macular degeneration) within 3 months of randomization.
* The subject is currently receiving dialysis.
* The subject is currently receiving or expected to require treatment (within the study period) with erythropoiesis medication such as epoetin alfa (Procrit, Epogen), or darbepoetin alfa (Aranesp).
* The subject has any of the following at screening:

Hemoglobin >15.5 gram (g)/decilitre (dL) (male subjects or post-menopausal females) Hemoglobin >14.5 g/dL (pre-menopausal female subjects) Single QTc >=480 millisecond (msec); or QTc >=500 msec in subjects with bundle branch block (these criteria do not apply to subjects with predominately paced rhythms) Aspartate aminotransferase and alanine aminotransferase >=2xupper limit of normal (ULN); alkaline phosphatase and bilirubin >=1.5xULN (isolated bilirubin >=1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) A positive pre-study drug/alcohol screen Lactation or pregnancy (as determined by positive serum or urine hCG test)

* The use of prohibited medications
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2014-10-08 (Actual); Study Completion 2014-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (13):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Canada (2):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Québec, Quebec

REFERENCES:
- [Derived] Aftab M, Coselli JS. Renal and visceral protection in thoracoabdominal aortic surgery. J Thorac Cardiovasc Surg. 2014 Dec;148(6):2963-6. doi: 10.1016/j.jtcvs.2014.06.072. Epub 2014 Jul 21. PMID 25135232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 10 centers in the United States and 2 centers in Canada from 31 October 2013 to 08 October 2014.
Pre-assignment Details: A total of 55 participants were randomized in the study and were included in All Subjects Population. Participants were stratified according to intervention type (surgical or endovascular repair, with the latter limited to 50% of the total study population).
Groups:
- GSK1278863 300 mg Loading + 100 mg QD: Eligible participants received GSK1278863 300 milligrams (mg) on Day -1 (12 +/- 4 hours prior to planned surgery) as a loading dose followed by GSK1278863 100 mg once daily (QD) for 4 days starting from Day 0 (surgical day).
- Placebo: Eligible participants received Placebo matching GSK1278863 300 mg on Day -1 (12 +/- 4 hours prior to planned surgery) as a loading dose followed by Placebo matching GSK1278863 100 mg QD for 4 days starting from Day 0 (surgical day).
Period: Overall Study
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Started | 27 | 28
Completed | 20 | 25
Not Completed | 7 | 3
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Recovery | 2 | 0
Not completed — Investigator discretion | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1278863 300 mg Loading + 100 mg QD: Eligible participants received GSK1278863 300 mg on Day -1 (12 +/- 4 hours prior to planned surgery) as a loading dose followed by GSK1278863 100 mg QD for 4 days starting from Day 0 (surgical day).
- Total: Total of all reporting groups
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Customized [Count of Participants; unit: Participants]
  21 to 88 years | 27 | 28 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 24 | 19 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Peak in Cerebrospinal Fluid (CSF) S100 Beta Within 48 Hours Following Descending Thoracic Aorta/Thoracoabdominal Aortic Aneurysm (DTA/TAAA) Repair
Description: S100 beta is a CSF biomarker that rise significantly in participants with neurologic injury following DTA/TAAA surgery. CSF samples were collected at Baseline and within 48 hours following DTA/TAAA repair to assess peak change from Baseline in CSF S100 beta. Baseline was defined at Day 0. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) to 48 hours following DTA/TAAA repair
Population: Pharmacodynamic (PD) population comprised of all participants from whom PD data was available. For the change from Baseline assessment, only those with both evaluable Baseline and post-dose values (so that the change could be calculated) were included in the analysis.
Measure: Mean (Standard Deviation); unit: Nanograms per liter (ng/L)
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 27
Nanograms per liter (ng/L) | 2748.19 (6212.035) | 566.78 (1897.172)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; Test type: Superiority; p = 0.0820, ANCOVA; Mean Difference (Final Values) = 2228.14, 95% CI 2-sided [-292.84 to 4749.11] — The point estimate was calculated as least square (LS) mean difference (final values) of S-100B Protein [test] and S-100B Protein [reference]

2. Primary Outcome: Change From Baseline to Peak in CSF Glial Fibrillary Acidic Protein (GFAP) Within 48 Hours Following DTA/TAAA Repair
Description: GFAP is a CSF biomarker that rise significantly in participants with neurologic injury following DTA/TAAA surgery. CSF samples for the analysis of GFAP was collected at Baseline and within 48 hours following DTA/TAAA repair to assess peak change from Baseline in CSF GFAP. Baseline was defined at Day 0. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) to 48 hours following DTA/TAAA repair
Population: PD population. For the change from Baseline assessment, only those with both evaluable Baseline and post-dose values (so that the change could be calculated) were included in the analysis.
Measure: Mean (Standard Deviation); unit: Microgram per liter (µg/L)
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 27
Microgram per liter (µg/L) | 1078.61 (2894.129) | 283.03 (1092.448)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; Test type: Superiority; p = 0.1997, ANCOVA; Mean Difference (Final Values) = 777.95, 95% CI 2-sided [-424.04 to 1979.94] — The point estimate was calculated as LS mean difference (final values) of GFAP [test] and GFAP [reference]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, considered to be medically significant or is associated with liver injury and impaired liver function.
Time Frame: Up to Follow-up (Day 45)
Population: All Subjects Population comprised of all participants who received at least one dose of study drug (GSK1278863 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  Any AEs | 26 | 23
  Any SAEs | 20 | 14

4. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance (PCI)
Description: Vital sign measurements included systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate. Criteria for vital sign values meeting PCI included: SBP < 70 millimeters of mercury (mmHg) and > 160 mmHg; DBP < 45 mmHg and > 110 mmHg. Data for participants with vital signs values outside the potential clinical importance range has been presented. Only those parameters for which at least one value of PCI was reported are summarized.
Time Frame: Up to Follow-up (Day 45)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  SBP | 2 | 1
  DBP | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Electrocardiography (ECG) Parameters
Description: Single 12-lead ECGs was obtained at each time point during the study using an ECG machine that automatically calculated the heart rate and measures PR, QRS, QT, and QT interval corrected for heart rate intervals. Data for participants with abnormal-clinical significant (CS) and abnormal-not clinically significant (NCS) ECG findings on post-operative Days 1, 2, 3, 4, 5, 6, 7 and during Follow-up Visits has been presented.
Time Frame: Up to Follow-up (Day 45)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  Post-operative Day 1, Abnormal-NCS: number analyzed (Participants) | 26 | 25
  Post-operative Day 1, Abnormal-NCS | 18 | 18
  Post-operative Day 2, Abnormal-NCS: number analyzed (Participants) | 24 | 24
  Post-operative Day 2, Abnormal-NCS | 18 | 17
  Post-operative Day 3, Abnormal-NCS: number analyzed (Participants) | 22 | 22
  Post-operative Day 3, Abnormal-NCS | 17 | 16
  Post-operative Day 3, Abnormal-CS: number analyzed (Participants) | 22 | 22
  Post-operative Day 3, Abnormal-CS | 1 | 1
  Post-operative Day 4, Abnormal-NCS: number analyzed (Participants) | 18 | 22
  Post-operative Day 4, Abnormal-NCS | 13 | 18
  Post-operative Day 5, Abnormal-NCS: number analyzed (Participants) | 17 | 21
  Post-operative Day 5, Abnormal-NCS | 14 | 17
  Post-operative Day 6, Abnormal-NCS: number analyzed (Participants) | 19 | 16
  Post-operative Day 6, Abnormal-NCS | 14 | 10
  Post-operative Day 7, Abnormal-NCS: number analyzed (Participants) | 22 | 22
  Post-operative Day 7, Abnormal-NCS | 15 | 15
  Follow-up, Abnormal-NCS: number analyzed (Participants) | 15 | 22
  Follow-up, Abnormal-NCS | 11 | 13

6. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters of PCI
Description: Blood samples for assessment of clinical chemistry parameters aspartate amino transferase (AST), alanine amino transferase (ALT), gamma glutamyl transferase (GGT), alkaline phosphatase, blood urea nitrogen (BUN), creatinine, glucose, sodium, creatine phosphokinase, potassium, chloride, total carbon dioxide, calcium, total and direct bilirubin, uric acid, albumin and total protein was done at Randomization, Day 0 (done prior to 100 mg on-call dosing), 1, 2, 3, 4, 5, 6 and 7. Only those parameters for which at least one value of PCI was reported are summarized. Data for participants with clinical chemistry values outside the PCI range has been presented.
Time Frame: Up to post-operative Day 7
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants | 19 | 18

7. Secondary Outcome: Number of Participants With Hematology Parameters of PCI
Description: Blood samples for assessment of hematology parameters platelet count, red blood cell count, white blood cell count, reticulocyte count, hemoglobin, hematocrit, mean corpuscle volume, mean corpuscle hemoglobin, mean corpuscle hemoglobin concentration, neutrophils, lymphocytes, monocytes, eosinophils and basophils was done at Randomization, Day 0 (done prior to 100 mg on-call dosing), 1, 2, 3, 4, 5, 6 and 7. Only those parameters for which at least one value of PCI was reported are summarized. Data for participants with hematology values outside the PCI range has been presented.
Time Frame: Up to post-operative Day 7
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants | 25 | 16

8. Secondary Outcome: Change From Baseline in Area Under Curve (AUC) for CSF S100 Beta to 48 Hours
Description: S100 beta was a CSF biomarker that rise significantly in participants with neurologic injury following DTA/TAAA surgery. AUC for CSF S100 beta from Baseline to 48 hours following DTA/TAAA repair was assessed to measure central nervous system injury. AUC was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Baseline was defined at Day 0. Change from Baseline was calculated as post-Baseline minus Baseline value.
Time Frame: Baseline(Day 0) to 48 hours following DTA/TAAA repair
Population: PD Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per liter (hour*ng/L)
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Hour*nanogram per liter (hour*ng/L) | 17263.25 (316.40) | 9758.27 (221.85)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; Test type: Superiority; p = 0.1530, ANOVA; Estimate of comparison (Ratio) = 1.77, 95% CI 2-sided [0.80 to 3.90] — The point estimate was calculated as Geometric mean ratio of S-100B[test] and S-100B[reference]

9. Secondary Outcome: Change From Baseline in AUC for CSF GFAP to 48 Hours
Description: GFAP was a CSF biomarker that rise significantly in participants with neurologic injury following DTA/TAAA surgery. AUC for CSF GFAP from Baseline to 48 hours following DTA/TAAA repair was assessed to measure central nervous system injury. AUC was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Baseline was defined at Day 0. Change from Baseline was calculated as post-Baseline minus Baseline value.
Time Frame: Baseline(Day 0) to 48 hours following DTA/TAAA repair
Population: PD Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per liter (hour*µg/L)
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Hour*microgram per liter (hour*µg/L) | 182.35 (15899.84) | 58.32 (1413.66)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; Test type: Superiority; p = 0.1377, ANOVA; Estimate of comparison (Ratio) = 3.13, 95% CI 2-sided [0.69 to 14.26] — The point estimate was calculated as Geometric mean ratio of GFAP[test] and GFAP[reference]

10. Secondary Outcome: Change From Baseline to Peak in CSF Biomarker Erythropoietin Within 48 Hours Following DTA/TAAA Repair
Description: CSF biomarker erythropoietin samples were collected for the analysis of ischemic neurologic injury. CSF samples were collected at Baseline and within 48 hours following DTA/TAAA repair to assess peak change from Baseline in CSF erythropoietin. Baseline was defined at Day 0. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) to 48 hours following DTA/TAAA repair
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 27
International units per liter (IU/L) | 1.34 (137.411) | 0.61 (1.582)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = 34.56, 95% CI 2-sided [21.95 to 47.17] — The point estimate was calculated as LS mean difference final values of Erythropoietin[test] and Erythropoietin[reference]

11. Secondary Outcome: Change From Baseline to Peak in CSF Biomarker Lactate Dehydrogenase Within 48 Hours Following DTA/TAAA Repair
Description: CSF biomarker lactate dehydrogenase samples were collected for the analysis of ischemic neurologic injury. CSF samples were collected at Baseline and within 48 hours following DTA/TAAA repair to assess peak change from Baseline in CSF lactate dehydrogenase. Baseline was defined at Day 0. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) to 48 hours following DTA/TAAA repair
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 27
Millimoles per liter (mmol/L) | 1.82 (2.021) | 1.28 (1.160)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; Test type: Superiority; p = 0.2404, ANCOVA; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [-0.37 to 1.45] — The point estimate was calculated as LS mean difference final values of Lactate Dehydrogenase[test] and Lactate Dehydrogenase[reference]

12. Secondary Outcome: Change From Baseline to Peak in CSF Biomarker Tau Protein Within 48 Hours Following DTA/TAAA Repair
Description: CSF biomarker tau protein samples were collected for the analysis of ischemic neurologic injury. CSF samples were collected at Baseline and within 48 hours following DTA/TAAA repair to assess peak change from Baseline in CSF tau protein. Baseline was defined at Day 0. Change from Baseline was calculated as post-Baseline minus Baseline value.
Time Frame: Baseline (Day 0) to 48 hours following DTA/TAAA repair
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 27
ng/L | 1729.25 (2177.526) | 751.21 (1053.951)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; Test type: Superiority; p = 0.0526, ANCOVA; Mean Difference (Final Values) = 925.88, 95% CI 2-sided [-10.73 to 1862.49] — The point estimate was calculated as LS mean difference final values of Tau Protein[test] and Tau Protein[reference]

13. Secondary Outcome: Change From Baseline to Peak in CSF Biomarker Neuron-specific Enolase (NSE) Within 48 Hours Following DTA/TAAA Repair
Description: CSF biomarker NSE samples were collected for the analysis of ischemic neurologic injury. CSF samples were collected at Baseline and within 48 hours following DTA/TAAA repair to assess peak change from Baseline in CSF NSE. Baseline was defined at Day 0. Change from Baseline was calculated as post-Baseline minus Baseline value.
Time Frame: Baseline (Day 0) to 48 hours following DTA/TAAA repair
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 27
µg/L | 9.31 (9.717) | 5.65 (7.214)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; Test type: Superiority; p = 0.0893, ANCOVA; Mean Difference (Final Values) = 4.11, 95% CI 2-sided [-0.65 to 8.87] — The point estimate was calculated as LS mean difference final values of Neuron Specific Enolase[test] and Neuron Specific Enolase[reference]

14. Secondary Outcome: Number of Participants With Neurologic Outcomes Assessed by the National Institutes of Health Stroke Scale (NIHSS)
Description: The NIHSS was a systematic assessment tool that provided a quantitative measure of stroke-related neurologic deficit. A trained observer rates the participant's ability to answer questions and perform activities. Ratings for each item are scored with 0 as normal, and there was an allowance for untestable items. The NIHSS scores were categorized as: No event (NIHSS score=0), Mild (NIHSS score 1-4), Moderate (NIHSS score 5-15), or Severe (NIHSS score >15). The single participant assessment required less than 10 minutes to complete. Data for participants with NIHSS administrated at surgical day, post-operative Day 1, Day 2, Day 7 and Follow-up Visit has been reported.
Time Frame: Surgical Day (Day 0), Post-operative Day 1, 2, 7 and follow-up (Day 45)
Population: PD population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  Surgical Day, No event (Score=0): number analyzed (Participants) | 27 | 26
  Surgical Day, No event (Score=0) | 27 | 23
  Surgical Day, Mild (Score 1-4): number analyzed (Participants) | 27 | 26
  Surgical Day, Mild (Score 1-4) | 0 | 3
  Post-operative Day 1, No event (Score=0): number analyzed (Participants) | 25 | 23
  Post-operative Day 1, No event (Score=0) | 11 | 14
  Post-operative Day 1, Mild (Score 1-4): number analyzed (Participants) | 25 | 23
  Post-operative Day 1, Mild (Score 1-4) | 4 | 7
  Post-operative Day 1, Moderate (Score 5-15): number analyzed (Participants) | 25 | 23
  Post-operative Day 1, Moderate (Score 5-15) | 4 | 1
  Post-operative Day 1, Severe (Score >15): number analyzed (Participants) | 25 | 23
  Post-operative Day 1, Severe (Score >15) | 6 | 1
  Post-operative Day 2, No event (Score=0): number analyzed (Participants) | 24 | 22
  Post-operative Day 2, No event (Score=0) | 11 | 15
  Post-operative Day 2, Mild (Score 1-4): number analyzed (Participants) | 24 | 22
  Post-operative Day 2, Mild (Score 1-4) | 4 | 3
  Post-operative Day 2, Moderate (Score 5-15): number analyzed (Participants) | 24 | 22
  Post-operative Day 2, Moderate (Score 5-15) | 3 | 3
  Post-operative Day 2, Severe (Score >15): number analyzed (Participants) | 24 | 22
  Post-operative Day 2, Severe (Score >15) | 6 | 1
  Post-operative Day 7, No event (Score=0): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, No event (Score=0) | 10 | 16
  Post-operative Day 7, Mild (Score 1-4): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Mild (Score 1-4) | 2 | 7
  Post-operative Day 7, Moderate (Score 5-15): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Moderate (Score 5-15) | 4 | 1
  Post-operative Day 7, Severe (Score >15): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Severe (Score >15) | 4 | 0
  Follow-up, No event (Score=0): number analyzed (Participants) | 18 | 25
  Follow-up, No event (Score=0) | 13 | 17
  Follow-up, Mild (Score 1-4): number analyzed (Participants) | 18 | 25
  Follow-up, Mild (Score 1-4) | 1 | 6
  Follow-up, Moderate (Score 5-15): number analyzed (Participants) | 18 | 25
  Follow-up, Moderate (Score 5-15) | 4 | 2

15. Secondary Outcome: Number of Participants With Neurologic Outcomes Assessed by Modified Rankin Scale (mRS)
Description: The mRS was a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The mRS was a 6 point disability scale with possible scores ranging from 0 up to 5. A separate category (of 6) was added for participants who died. The mRS scores were categorized as mild (mRS score 0-1), moderate (mRS score 2-3), or severe (mRS score >=4).
Time Frame: Post-operative Day 7 and follow-up (Day 45)
Population: PD population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  Post-operative Day 7, Mild (Score 0-1): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Mild (Score 0-1) | 9 | 11
  Post-operative Day 7, Moderate (Score 2-3): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Moderate (Score 2-3) | 1 | 8
  Post-operative Day 7, Severe (Score >=4): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Severe (Score >=4) | 10 | 5
  Follow-up, Mild (Score 0-1): number analyzed (Participants) | 18 | 25
  Follow-up, Mild (Score 0-1) | 8 | 14
  Follow-up, Moderate (Score 2-3): number analyzed (Participants) | 18 | 25
  Follow-up, Moderate (Score 2-3) | 4 | 7
  Follow-up, Severe (Score >=4): number analyzed (Participants) | 18 | 25
  Follow-up, Severe (Score >=4) | 6 | 4

16. Secondary Outcome: Number of Participants With Neurologic Outcomes Assessed by the American Spinal Injury Association (ASIA) Lower Extremity Motor Outcome Scale
Description: The ASIA score was developed by the American Spinal Injury Association for the neurologic assessment of participants with a spinal injury. In this study, only the ASIA lower extremity motor score was assessed. This comprised five muscle groups scored from 0-5 on both the left and right lower extremities, for a maximal total score of 50. The ASIA scores were categorized as: mild (ASIA score 41-50), moderate (ASIA score 26-40), or severe (ASIA score <=25).
Time Frame: Surgical Day (Day 0), Post-operative Day 1, 2, 7 and follow-up (Day 45)
Population: PD population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  Surgical Day, Mild (Score 41-50): number analyzed (Participants) | 27 | 26
  Surgical Day, Mild (Score 41-50) | 26 | 26
  Surgical Day, Moderate (Score 26-40): number analyzed (Participants) | 27 | 26
  Surgical Day, Moderate (Score 26-40) | 1 | 0
  Post-operative Day 1, Mild (Score 41-50): number analyzed (Participants) | 25 | 23
  Post-operative Day 1, Mild (Score 41-50) | 15 | 19
  Post-operative Day 1, Moderate (Score 26-40): number analyzed (Participants) | 25 | 23
  Post-operative Day 1, Moderate (Score 26-40) | 2 | 2
  Post-operative Day 1, Severe (Score <=25): number analyzed (Participants) | 25 | 23
  Post-operative Day 1, Severe (Score <=25) | 8 | 2
  Post-operative Day 2, Mild (Score 41-50): number analyzed (Participants) | 23 | 22
  Post-operative Day 2, Mild (Score 41-50) | 14 | 21
  Post-operative Day 2, Moderate (Score 26-40): number analyzed (Participants) | 23 | 22
  Post-operative Day 2, Moderate (Score 26-40) | 1 | 0
  Post-operative Day 2, Severe (Score <=25): number analyzed (Participants) | 23 | 22
  Post-operative Day 2, Severe (Score <=25) | 8 | 1
  Post-operative Day 7, Mild (Score 41-50): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Mild (Score 41-50) | 13 | 22
  Post-operative Day 7, Moderate (Score 26-40): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Moderate (Score 26-40) | 1 | 1
  Post-operative Day 7, Severe (Score <=25): number analyzed (Participants) | 20 | 24
  Post-operative Day 7, Severe (Score <=25) | 6 | 1
  Follow-up, Mild (Score 41-50): number analyzed (Participants) | 18 | 25
  Follow-up, Mild (Score 41-50) | 14 | 24
  Follow-up, Moderate (Score 26-40): number analyzed (Participants) | 18 | 25
  Follow-up, Moderate (Score 26-40) | 2 | 0
  Follow-up, Severe (Score <=25): number analyzed (Participants) | 18 | 25
  Follow-up, Severe (Score <=25) | 2 | 1

17. Secondary Outcome: Number of Participants With Clinical Composite of All Cause Mortality, Stroke, Spinal Infarction, MI, Need for Dialysis/Sustained Doubling of Serum Creatinine
Description: The clinical composite event rate included all-cause mortality (death), stroke, spinal infarction (paraplegia which was due to spinal infarct a result of the surgery, myocardial infarction, and the need for dialysis or sustained doubling of serum creatinine (acute kidney injury). The clinical composite endpoint used a first occurrence approach, i.e. a composite event was recorded at the time of first occurrence of any component of the composite.
Time Frame: Up to Follow-up (Day 45)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  Acute Kidney Injury | 13 | 10
  Myocardial Infarction | 1 | 0
  Paraplegia | 6 | 4
  Stroke | 1 | 2
  Death | 6 | 2
  Composite Above | 16 | 12

18. Secondary Outcome: Assessment in AUC for Markers of Ischemic Organ Injury Including Tropinin Within 48 Hours
Description: AUC from 8 hours post surgery (up to 48 hours post surgery) was derived for markers of ischemic organ injury troponin I and troponin T. AUC was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: Baseline (Day 0) and 8 to 48 hours following DTA/TAAA repair
Population: PD population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hour/L
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
µg*hour/L
  Troponin I: number analyzed (Participants) | 19 | 17
  Troponin I | 13.29 (0.615) | 7.23 (0.650)
  Troponin T: number analyzed (Participants) | 8 | 11
  Troponin T | 3.14 (0.879) | 4.19 (0.750)
Statistical Analysis 1: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; For Troponin I; Test type: Superiority; p = 0.5012, ANOVA; Ratio of geometric mean = 1.84, 95% CI 2-sided [0.30 to 11.32]
Statistical Analysis 2: Comparison: GSK1278863 300 mg Loading + 100 mg QD vs Placebo; For Troponin T; Test type: Superiority; p = 0.8053, ANOVA; Ratio of geometric mean = 0.75, 95% CI 2-sided [0.07 to 8.57]

19. Secondary Outcome: Number of Participants With Composite Index of All Cause Mortality and Disability (NIHSS>5/ASIA<40)
Description: The NIHSS was a systematic assessment tool that provided a quantitative measure of stroke-related neurologic deficit. Ratings for each item are scored with 0 as normal, and there was an allowance for untestable items. The NIHSS scores were categorized as: No event (NIHSS score=0), Mild (NIHSS score 1-4), Moderate (NIHSS score 5-15), or Severe (NIHSS score >15). The ASIA score was developed by the American Spinal Injury Association for the neurologic assessment of participants with a spinal injury. In this study, only the ASIA lower extremity motor score was assessed. This comprised five muscle groups scored from 0-5 on both the left and right lower extremities, for a maximal total score of 50. The ASIA scores were categorized as: mild (ASIA score 41-50), moderate (ASIA score 26-40), or severe (ASIA score <=25). "Composite above" includes participants with NIHSS>5 or ASIA<40 at the 30-day Follow-up or Death.
Time Frame: Up to Follow-up (Day 45)
Population: PD Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  ASIA <40 | 4 | 1
  NIHSS >5 | 4 | 2
  Death | 6 | 2
  Composite Above | 11 | 4

20. Secondary Outcome: Pharmacokinetic (PK) Parameters in Blood: AUC(0-t) of GSK1278863
Description: Blood samples for PK analysis AUC(0-t) were collected at pre-dose (prior to the 100 mg dose), 1-3 hours after study drug was administered and then every 5 hours for 24 hours. On Days 1 and 3 samples were collected at pre-dose then 1, 3, 8 and 24 hours post dose. AUC (0-t) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: Pre-dose, 1 to 3 hours post-dose, every 5 hours for 24 hours, 1, 3, 8 and 24 hours post-dose on Day 1 and 3
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*ng/mL
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD
Number analyzed (Participants) | 27
Hour*ng/mL
  Blood, Surgical Day: number analyzed (Participants) | 26
  Blood, Surgical Day | 3591.449 (50.23)
  Blood, Post-operative Day 1 | 2858.165 (129.26)
  Blood, Post-operative Day 3: number analyzed (Participants) | 23
  Blood, Post-operative Day 3 | 3710.790 (115.20)

21. Secondary Outcome: PK Parameters in CSF: AUC(0-t) of GSK1278863
Description: CSF samples were collected immediately after the lumbar drain was placed, just prior to PNI, and 2, 24, 36 and 48 hours post PNI. In participants that developed spinal ischemia, the CSF drain was potentially maintained for longer than 48 hours. In that instance, daily CSF samples for PK were collected until the drain was removed. AUC (0-t) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: Prior to potential neurological ischemia (PNI), 2, 24, 36 and 48 hours post PNI
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*ng/mL
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD
Number analyzed (Participants) | 26
Hour*ng/mL | 37.340 (156.10)

22. Secondary Outcome: PK Parameters in Blood: Maximum Observed Concentration (Cmax) of GSK1278863
Description: as for outcome 20
Time Frame: Pre-dose, 1 to 3 hours post-dose, every 5 hours for 24 hours, 1, 3, 8 and 24 hours post-dose on Day 1 and 3
Population: PK population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ng/mL
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD
Number analyzed (Participants) | 27
Ng/mL
  Blood, Surgical Day: number analyzed (Participants) | 26
  Blood, Surgical Day | 705.701 (83.43)
  Blood, Post-operative Day 1 | 358.518 (192.32)
  Blood, Post-operative Day 3: number analyzed (Participants) | 23
  Blood, Post-operative Day 3 | 779.801 (110.20)

23. Secondary Outcome: PK Parameters in CSF: Cmax of GSK1278863
Description: as for outcome 21
Time Frame: Prior to potential neurological ischemia (PNI), 2, 24, 36 and 48 hours post PNI
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ng/L
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD
Number analyzed (Participants) | 26
Ng/L | 2.364 (105.24)

24. Secondary Outcome: PK Parameters in Blood: Time of Occurrence of Cmax (Tmax) of GSK1278863
Description: as for outcome 20
Time Frame: Pre-dose, 1 to 3 hours post-dose, every 5 hours for 24 hours, 1, 3, 8 and 24 hours post-dose on Day 1 and 3
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD
Number analyzed (Participants) | 27
Hours
  Blood, Surgical day: number analyzed (Participants) | 26
  Blood, Surgical day | 1.725 [0.00 to 16.38]
  Blood, Post-operative Day 1 | 3.017 [0.02 to 24.43]
  Blood, Post-operative Day 3: number analyzed (Participants) | 23
  Blood, Post-operative Day 3 | 3.017 [0.77 to 8.18]

25. Secondary Outcome: PK Parameters in CSF: Tmax of GSK1278863
Description: as for outcome 21
Time Frame: Prior to potential neurological ischemia (PNI), 2, 24, 36 and 48 hours post PNI
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD
Number analyzed (Participants) | 26
Hours | 15.326 [8.097 to 22.554]

ADVERSE EVENTS:
Time Frame: AEs were collected up to Follow-up (Day 45).
Description: All Subjects Population was used.
Arm/Group | GSK1278863 300 mg Loading + 100 mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 6/27 | 2/28
Serious Adverse Events (participants affected / at risk) | 20/27 | 14/28
Other Adverse Events (participants affected / at risk) | 20/27 | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1278863 300 mg Loading + 100 mg QD (N=27) | Placebo (N=28)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Spinal cord ischaemia (Nervous system disorders) | 2 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 4 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Haemodynamic instability (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 5 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 2 | 0
Internal injury (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Cystitis klebsiella (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Multi-organ failure (General disorders) | 4 | 0
Ischaemic ulcer (General disorders) | 1 | 0
Pulse absent (Investigations) | 1 | 0
Red blood cells CSF positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1278863 300 mg Loading + 100 mg QD (N=27) | Placebo (N=28)
Hypertension (Vascular disorders) | 3 | 6
Hypotension (Vascular disorders) | 4 | 5
Ischaemia (Vascular disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Coagulopathy (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 3
Bradycardia (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 5
Vomiting (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 4 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 3
Wound complication (Injury, poisoning and procedural complications) | 2 | 2
Headache (Nervous system disorders) | 3 | 4
Vocal cord paralysis (Nervous system disorders) | 1 | 2
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 2 | 1
Catheter site pain (General disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 3
Respiratory tract infection (Infections and infestations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Anxiety (Psychiatric disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 2
Troponin increased (Investigations) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.